CLINICAL TRIAL: NCT00965627
Title: Biological Analysis of a Series of Thymoma and Thymic Carcinoma: Genetic Aberrations and Potential Therapy Targets.
Brief Title: Biology of Thymic Tumors
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Armando Santoro, MD, Istituto Clinico Humanitas
Other Study IDs: ONC/OSS-01/2008
Record Dates: First submitted 2009-08-06; First posted 2009-08-25 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2009-08

CONDITIONS: Thymoma
MeSH Terms: conditions — Thymoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — paraffin-embedded tumor specimens of patients
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective analysis of biological characteristics of thymoma and thymic carcinoma patients.

DETAILED DESCRIPTION:
The aim of the present study is to investigated the genetic alterations in tumor samples of a series of all WHO-defined subtypes of thymoma patients using high resolution microarray- comparative genomic hybridization (CGH) followed by hierarchical cluster analyses of the data to identify specific patterns of genetic aberrations and genes associated with each subtype. Moreover, tumor samples will be also investigated for some specific potential therapy targets by immunoistichemistry, mutation analysis, and fluorescence in situ hybridization (FISH) analysis. All these biological data will be correlated with clinical patients characteristics and survival data.

ELIGIBILITY:
Inclusion Criteria:

* Availability of tumor tissue and patients with thymoma and thymic carcinoma

Exclusion Criteria:

* NON Availability of tumor tissue and patients with thymoma and thymic carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thymoma and thymic carcinoma patients will be retrospectively analyzed. Patients will be selected based on the availability of tumor tissue.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2008-06; Primary Completion 2008-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Primary objective: to evaluate the presence of genetic alterations and specific potential therapy targets. | one year

SECONDARY OUTCOMES:
Secondary objective: to correlate the biological characteristics with clinical characteristics and survival data of patients. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

REFERENCES:
- [Derived] Petrini I, Wang Y, Zucali PA, Lee HS, Pham T, Voeller D, Meltzer PS, Giaccone G. Copy number aberrations of genes regulating normal thymus development in thymic epithelial tumors. Clin Cancer Res. 2013 Apr 15;19(8):1960-71. doi: 10.1158/1078-0432.CCR-12-3260. Epub 2013 Feb 26. PMID 23444221